CLINICAL TRIAL: NCT00866749
Title: Augmented Berlin-Frankfurt-Munster Therapy for Adolescents/Young Adults With Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Brief Title: Augmented Berlin-Frankfurt-Munster (BFM) Therapy for Adolescent/Young Adults With Acute Lymphoblastic Leukemia or Acute Lymphoblastic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0375; NCI-2012-01650 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: acute lymphoblastic leukemia; acute lymphoblastic lymphoma; Leukemia; ALL; 6-Thioguanine; Cyclophosphamide; Cytarabine; Daunorubicin; Doxorubicin; Methotrexate; PEG-L-Asparaginase; Vincristine; Intrathecal Methotrexate; Mercaptopurine
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Daunorubicin; Vincristine; pegaspargase; Methotrexate; Cyclophosphamide; Cytarabine; Mercaptopurine; Doxorubicin; Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Augmented BFM Therapy (Experimental): Induction + Maintenance: Daunorubicin, Vincristine, PEG-asparaginase, Intrathecal Methotrexate, Cyclophosphamide, Cytarabine, Mercaptopurine, Doxorubicin, Thioguanine
  Interventions: Drug: Daunorubicin; Drug: Vincristine; Drug: PEG-asparaginase; Drug: Intrathecal Methotrexate; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Doxorubicin; Drug: Thioguanine

INTERVENTIONS:
Drug: Daunorubicin — Starting Dose 25 mg/m^2 by vein weekly
  Other Names: Cerubidine®
Drug: Vincristine — Starting Dose 2 mg by vein weekly
  Other Names: Vincasar®
Drug: PEG-asparaginase — Starting Dose 2000 International units/m2 by vein in week 1
  Other Names: Oncaspar®
Drug: Intrathecal Methotrexate — Starting Dose 12 mg on week 2 and week 5 injected into spinal fluid
  Other Names: Rheumatrex®
Drug: Cyclophosphamide — Starting Dose 1g/m2 by vein in weeks 1 and 5
  Other Names: Cytoxan®
Drug: Cytarabine — 75 mg/m2 subcutaneous or by vein for four consecutive days on days 1-4 and days 8-11 of both months
  Other Names: Cytosar-U®
Drug: Mercaptopurine — Starting Dose 60 mg/m2 by mouth on days 1-14 of each month
  Other Names: Purinethol®
Drug: Methotrexate — Starting Dose at 100 mg/m2 by vein and escalating by 50 mg/m2/dose every 10
  +/- 2 days for 5 doses to toxicity (e.g myelosuppression or mucositis grade 3
  Other Names: Rheumatrex®
Drug: Doxorubicin — 25 mg/m2 by vein in weeks 1, 2 and 3
  Other Names: Adriamycin®
Drug: Thioguanine — 60 mg/m2 by mouth daily for two weeks
  Other Names: Thioguanine Tabloid®

SUMMARY:
Objectives:

A. Primary objective:

1 To assess the feasibility and the effectiveness of pediatric type therapy (augmented BFM) in patients age 12 through 40 with untreated precursor-B or T acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LL).

B. Secondary objective:

1. To evaluate the prognostic significance of minimal residual disease in bone marrow samples at the end of induction and at the end of consolidation in this group of patients.
2. To prospectively evaluate gene hypermethylation status in this group of patients.
3. To prospectively analyze asparaginase activity and anti-asparaginase antibody formation in this population of patients.

DETAILED DESCRIPTION:
Induction:

During Induction, you will receive augmented Berlin-Frankfurt-Munster chemotherapy, which is made up of a combination of Cerubidine®, Daunorubicin Hydrochloride (daunorubicin), Oncovin® (vincristine), prednisone, dexamethasone, Oncaspar® (PEG Asparaginase), and MTX amethopterin (methotrexate). All of these drugs are designed to interfere with the multiplication of cancer cells to cause them to die and to keep the cancer from coming back.

If you are found to be eligible to take part in this study, on Day 1 or during the spinal tap procedure, you will be given cytarabine as an injection in your spinal fluid. Within 3 days, you will begin the Induction course, which will last for 4 weeks.

Daunorubicin and vincristine will be given through a needle in your vein on Days 1, 8,15, and 22. During the first week of therapy, you will be given 1 infusion of PEG Asparaginase by vein. You will take prednisone by mouth on Days 1-28. Methotrexate will be injected into your spinal fluid on Weeks 2 and 5 during your spinal tap. Cerebrospinal fluid (CSF) studies will be sent with each spinal tap to test the fluid for leukemia. If there is disease in your spinal fluid before starting the treatment, you will be given additional methotrexate doses once a week until there is no disease present. You will continue to receive methotrexate in spinal taps every other week for 8 doses, then monthly for 6 doses.

Blood (about 3 teaspoons) will be drawn multiple times during the study for routine tests. You will have a bone marrow aspirate or biopsy on Days 15 and 29 and then as needed to confirm remission.

If you have less than 5% immature cells in the bone marrow, 1 week after Induction, you will continue treatment with Consolidation 1. If you achieved remission after 4 weeks of Induction treatment, you will then have treatment with Consolidation 1, which will be discussed in a separate informed consent document.

If you have LL and had no bone marrow involvement at screening, you will have a chest x-ray, CT scans, and PET scans to measure the disease. Consolidation 1 and other phases of chemotherapy will be discussed in a separate informed consent document.

If you still have more than 5% leukemia cells in the bone marrow after Induction therapy, you will receive 2 extra weeks of therapy called "Extended Induction" before going to the next phase of therapy. You will receive daunorubicin by vein on Day 1. You will receive vincristine on Weeks 1 and 2 by vein. You will take prednisone by mouth on Days 1-14. You will receive PEG Asparaginase by vein in the first week of the Extended Induction. Blood (about 3 teaspoons) will be drawn weekly during the Extended Induction period for routine tests.

At the end of the Extended Induction period, you will have a physical exam and a bone marrow aspirate or biopsy to learn your response to treatment.

After Extended Induction, if the disease is in remission, then you will have 1 course of Consolidation 1, 2 courses of Consolidation 2, and 2 courses of Consolidation 3 before proceeding to Maintenance therapy. A separate discussion and informed consent document for Consolidation and Maintenance will be provided.

Length of Study:

You may remain on study for as long as you are benefiting. However, if after Extended Induction, the disease is not in remission, you will be taken off study, and your doctor will discuss other treatment options with you.

You may be taken off study if the disease gets worse or comes back during treatment, intolerable side effects occur, new information becomes available to your study doctor, if your doctor thinks it is in your best interest, or if you do not attend your appointments, which are scheduled at least once every 3 months.

This is an investigational study. The chemotherapy drugs used in this study are FDA approved and commercially available. Up to 125 patients will take part in this study. All will be enrolled at MD Anderson.

Consolidation and Maintenance:

During Consolidation, you will receive cyclophosphamide, cytarabine, 6-mercaptopurine, vincristine, PEG asparaginase, methotrexate, doxorubicin, 6-thioguanine, and dexamethasone. During Maintenance, you will receive, vincristine, dexamethasone, 6-mercaptopurine, and methotrexate. All of these drugs are designed to interfere with the multiplication of cancer cells to cause them to die and to keep the cancer from coming back.

If you achieved remission after 4 weeks of induction treatment, you will have treatment with Consolidation 1, Consolidation 2, Consolidation 3 (Parts A and B), and then you will proceed to Maintenance therapy.

If the level of blast cells in your blood is above a certain level at Day 15 of Induction but you achieved complete remission by Day 29, or if you achieved remission after 6 weeks of induction plus extended induction, then you will receive 1 course of Consolidation 1, 2 courses of Consolidation 2, 2 courses of Consolidation 3 (Parts A and B), and then you will proceed to maintenance therapy.

Consolidation 1 will last for 8 weeks (2 months). You will receive cyclophosphamide through a needle in your vein on Weeks 1 and 5. Cytarabine will be given as an injection just beneath the skin or by vein on or around Days 1-4 and Days 8-11 of each month. 6-Mercaptopurine will be taken by mouth on Days 1-14 of each month. Vincristine will be given by vein on Weeks 3-4 of each month. PEG Asparaginase will be given by vein on Week 3 and 6 of each month. You will receive methotrexate through a needle through your spine weekly during Month 1 only. Blood (about 3 teaspoons) will be drawn for routine tests. You will have a spinal tap with spinal fluid tests during the intrathecal methotrexate dose. A spinal tap (also called a lumbar puncture) is when a special needle is inserted into the lower back through the space between the bones to draw a sample of the fluid that surrounds the spinal cord. You will have a bone marrow aspiration at the end of Month 2. To collect a bone marrow aspirate, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

Consolidation 2 will last for 7 weeks. You will receive vincristine and methotrexate by vein every 10 plus or minus 2 days for 5 doses. You will receive PEG Asparaginase by vein in Weeks 1 and 4. You will receive intrathecal methotrexate in Weeks 1 and 5. You will have a spinal tap with spinal fluid tests during the intrathecal methotrexate dose. Blood (about 3 teaspoons) will be drawn every 2 weeks for routine tests.

Consolidation 3 (Part A) will last for 4 weeks. You will receive vincristine and Doxorubicin by vein in Weeks 1, 2 and 3. Dexamethasone will be taken by mouth on Days 1-7 and Days 15-21. You will receive PEG Asparaginase by vein on Week 1. You will receive intrathecal methotrexate in Week 1.

Consolidation 3 (Part B) will last for 4 weeks. You will receive cyclophosphamide by vein in Week 1. You will receive cytarabine by vein or as an injection for 4 days in a row in Weeks 1-2. You will take 6-Thioguanine by mouth every day for the first 2 weeks. You will receive intrathecal methotrexate in Weeks 1 and 2. You will receive vincristine by vein on Weeks 3 and 4. You will receive PEG Asparaginase by vein on Week 3.

During Consolidation 3 (Part A and B), blood (about 3 teaspoons) will be drawn at least weekly for routine tests. Spinal fluid tests will be sent with each intrathecal methotrexate dose. Spinal taps will be done during each intrathecal chemotherapy dose

Once you finish Consolidation, you will proceed to maintenance therapy.

The Maintenance period for ALL patients will last for 24 months. If you have ALL, you will receive vincristine by vein every month. You will take dexamethasone by mouth for 5 days every month. You will take 6-Mercaptopurine by mouth once daily. You will take methotrexate by mouth every week. You will receive intrathecal methotrexate every 3 months for the first 12 months of maintenance. You will have a spinal tap with spinal fluid tests during the intrathecal methotrexate dose.

Maintenance for patients with LL will also last for 24 months. If you have LL, you will receive vincristine by vein every month. You will take dexamethasone by mouth for 5 days every month.

You will take 6-Mercaptopurine by mouth once daily. You will take methotrexate by mouth every week.

During the Maintenance period, all participants will have blood samples (about 1 to 3 teaspoons each time) drawn every 3 months for routine tests.

If you have LL, you will have an additional positron emission tomography (PET) scan and computed tomography (CT) scan at the end of the Maintenance period.

Follow-Up Visits:

Your study doctor will inform you of your follow-up visits in the clinic. At each follow-up visit there will be a physical exam and complete blood count. You will be followed-up for the next 3 years after your the last dose of your chemotherapy.

Length of Study:

You may remain on study for as long as you are benefiting. You may be taken off study if the disease gets worse or comes back during treatment, intolerable side effects occur, new information becomes available to your study doctor, if your doctor thinks it is in your best interest, or if you do not attend your appointments, which are scheduled at least once every 3 months.

This is an investigational study. The chemotherapy drugs used in this study are all FDA approved and commercially available. Up to 125 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have precursor-B or T-lymphoblastic leukemia or lymphoblastic lymphoma.
2. Patients must be untreated or have had only one prior chemotherapy regimen for ALL or LL . Previously treated patients will be analyzed separately.
3. Age between 12 to 40 years old
4. Patients with Central Nervous System (CNS) disease or testicular disease are eligible.
5. Intrathecal therapy with cytarabine is allowed prior to registration for patient convenience. This is usually done at the time of the diagnostic bone marrow or venous line placement to avoid a second lumbar puncture. Systemic chemotherapy must begin within 72 hours of the first intrathecal treatment.
6. Signed informed consent prior to the start of systemic therapy. In the event of enrollment of a minor patient, an attempt to obtain assent from the patient must be documented, and parental consent must be signed.
7. Echocardiogram should be done within 72 hours of starting therapy if there are cardiac risk factors (e.g., history of hypertension or of myocardial infarction)
8. Creatinine should be < 3 mg/dL bilirubin < 3 mg/dl unless felt to be due to disease
9. Zubrod Performance status of <3
10. Patients who received steroids more than 72 hours prior to study enrollment are eligible but will be analyzed separately

Exclusion Criteria:

1. Age less than twelve years of age or greater than 40 years.
2. More than one prior treatment regimen for ALL or LL.
3. The patient is pregnant or unwilling to practice appropriate birth control.
4. Presence of the Philadelphia chromosome t(9;22)

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2006-09-12 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E. Rytting, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 2006 - March 2014
Groups:
- Augmented BFM Therapy: Induction + Maintenance: Daunorubicin, Vincristine, PEG-asparaginase, Intrathecal Methotrexate, Cyclophosphamide, Cytarabine, Mercaptopurine, Doxorubicin, Thioguanine
  Daunorubicin: Starting Dose 25 mg/m^2 by vein weekly
  Vincristine: Starting Dose 2 mg by vein weekly
  PEG-asparaginase: Starting Dose 2000 International units/m2 by vein in week 1
  Intrathecal Methotrexate: Starting Dose 12 mg on week 2 and week 5 injected into spinal fluid
  Cyclophosphamide: Starting Dose 1g/m2 by vein in weeks 1 and 5
  Cytarabine: 75 mg/m2 subcutaneous or by vein for four consecutive days on days 1-4 and days 8-11 of both months
  Mercaptopurine: Starting Dose 60 mg/m2 by mouth on days 1-14 of each month
  Methotrexate: Starting Dose at 100 mg/m2 by vein and escalating by 50 mg/m2/dose every 10
  +/- 2 days for 5 doses to toxicity (e.g myelosuppression or mucositis grade 3
  Doxorubicin: 25 mg/m2 by vein in weeks 1, 2 and 3
  Thioguanine: 60 mg/m2 by mouth daily for two weeks
Period: Overall Study
Arm/Group | Augmented BFM Therapy
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Augmented BFM Therapy
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24
  Between 18 and 65 years | 96
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 22 [13 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 104
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 120

OUTCOME MEASURES:

1. Primary Outcome: 3-Year Event-Free Survival (EFS)
Description: 3-year EFS was calculated based on the participants with a complete response (CR). Study regimen considered successful if it exhibits a 3-year EFS rate greater than 60% and response rate no less than 90% with Grade III-IV infectious toxicity rate in induction no more than 33%.
Time Frame: 3 Years
Population: Of the 108 participants who had a complete response, 68 met the definition for 3 year EFS.
Measure: Count of Participants; unit: Participants
Arm/Group | Augmented BFM Therapy
Number analyzed (Participants) | 108
Participants | 68

2. Primary Outcome: Overall Survival
Description: Overall Survival defined: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 12 years
Measure: Median (Full Range); unit: Months
Arm/Group | Augmented BFM Therapy
Number analyzed (Participants) | 120
Months | 121 [0.5 to 140]

3. Primary Outcome: Participants With a Complete Response (CR)
Description: Complete Response defined as: Bone Marrow blasts </= 5%, Platelets >/= 100 and an Absolute Neutrophil Count (ANC) >/= 1000
Time Frame: Up to 1 year
Measure: Number; unit: participants
Arm/Group | Augmented BFM Therapy
Number analyzed (Participants) | 120
participants | 108

4. Secondary Outcome: Participants Achieving Negative Minimal Residual Disease (MRD)
Description: To evaluate the prognostic significance of minimal residual disease (MRD) in bone marrow samples of participants who achieved a complete response (CR) at the end of induction (day 29) and at the end of consolidation (day 84) in this group of patients.
Time Frame: up to 3 months
Population: Of the 108 participants who achieved a complete response (CR), 60 participants were MRD negative on day 29 and an additional 27 participants were MRD negative on day 84 for a total 87 MRD negative participants on day 84
Measure: Number; unit: participants
Arm/Group | Augmented BFM Therapy
Number analyzed (Participants) | 108
participants
  Participants with CR and MRD negative on Day 29 | 60
  Participants with CR and MRD negative on day 84 | 87

ADVERSE EVENTS:
Time Frame: Participants were assessed through study completion, for up to 3 years.
Arm/Group | Augmented BFM Therapy
All-Cause Mortality (participants affected / at risk) | 6/120
Serious Adverse Events (participants affected / at risk) | 64/120
Other Adverse Events (participants affected / at risk) | 111/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Augmented BFM Therapy (N=120)
Abdominal Cramps (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 7 (15)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Ankle Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety/depression (Psychiatric disorders) | 2 (2)
Avascular Necrosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone Pain (General disorders) | 1 (1)
Central Nervous System, White matter (Nervous system disorders) | 1 (1)
Cerebrovascular Ischemia (Nervous system disorders) | 1 (1)
Cognitive Disturbance (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cytomegalovirus antigen positive (General disorders) | 2 (3)
Dehydration (Gastrointestinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Double vision (Eye disorders) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Elevated Alanine Aminotransferase (Investigations) | 1 (1)
Embolism (Vascular disorders) | 3 (3)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 11 (16)
Gallbladder Obstruction (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Generalized Edema (General disorders) | 1 (1)
Groin Abscess (General disorders) | 1 (1)
Headache (General disorders) | 7 (10)
Hemorrhage (General disorders) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 3 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 22 (29)
Knee Pain (General disorders) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 6 (6)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 5 (6)
Neuropathy (Nervous system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenic Fever (Infections and infestations) | 30 (51)
Osteoprosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 7 (9)
Pleuritic Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Pulmonary Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Syncytial Virus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Striae (Skin and subcutaneous tissue disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1)
Vaginal Herpes (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Augmented BFM Therapy (N=120)
Colitis (Gastrointestinal disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Supraventricualr arrhythmia (Cardiac disorders) | 6 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (9)
Dehydration (Gastrointestinal disorders) | 9 (9)
Lipase (Metabolism and nutrition disorders) | 9 (9)
Mucositis (Gastrointestinal disorders) | 22 (26)
Constipation (Gastrointestinal disorders) | 11 (11)
Pain (General disorders) | 29 (38)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 11 (12)
Pancreatitis (Gastrointestinal disorders) | 11 (12)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 13 (13)
Neutropenic Fever (Infections and infestations) | 12 (15)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 15 (15)
Neuropathy motor (Nervous system disorders) | 19 (21)
Nausea (Gastrointestinal disorders) | 19 (23)
Hyperglycemia (Metabolism and nutrition disorders) | 22 (24)
Neuropathy sensor (Nervous system disorders) | 23 (24)
Allergic reaction/hypersensitivity (Immune system disorders) | 23 (25)
Thrombosis (Vascular disorders) | 22 (29)
Infection (Infections and infestations) | 70 (138)
Fibrinogen (Investigations) | 43 (44)
Elevated Alanine Aminotransferase (Investigations) | 25 (78)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 57 (87)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT00866749/Prot_SAP_000.pdf